CLINICAL TRIAL: NCT00358358
Title: A Randomized, Double-blind Placebo-controlled Study of Treatments With Salmeterol, Fluticasone Propionate and Their Combination to Evaluate Novel Endpoints in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Chronic Obstructive Pulmonary Disease Endpoints Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCO104925
Record Dates: First submitted 2006-07-27; First posted 2006-07-31 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; Impulse Oscillometry System; Computerized Tomography
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone; Salmeterol Xinafoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Fluticasone Propionate/Salmeterol 500/50mcg combination
Drug: Fluticasone Propionate 500mcg
Drug: Salmeterol 50mcg
  Other Names: Fluticasone Propionate/Salmeterol 500/50mcg combination; Fluticasone Propionate 500mcg

SUMMARY:
This study will last for approximately 14 weeks and will involve 5 visits. The study is being carried out to look at different ways of measuring the effect of drug treatment on COPD. COPD is a respiratory disease which can affect your breathing and daily life. Symptoms of COPD can include breathlessness, cough, and wheeze. COPD varies enormously from patient to patient. The effects of drug treatment are usually measured by conducting lung function tests (breathing tests) using a machine called a spirometer but this does not always provide a complete picture of how well your COPD is responding. In this study we therefore want to look at new and more sensitive ways of measuring COPD. The results of this research will help in the assessment of new drugs for COPD in the future.

DETAILED DESCRIPTION:
Evaluation of Novel Endpoints in Subjects with Chronic Obstructive Pulmonary Disease (COPD) in a Randomized, Double-Blind, Placebo-Controlled Study of Treatment with Fluticasone Propionate/Salmeterol 500/50mcg combination (FSC 500/50) and its individual components, Fluticasone Propionate 500mcg (FP500) and Salmeterol 50mcg (SAL 50)

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of COPD
* Current or ex-smoker at least 10 pack- years

Exclusion criteria:

* Diagnosis of asthma
* Active respiratory disorder other than COPD
* Evidence of clinically significant uncontrolled non-pulmonary disease
* Carcinoma not in complete remission for last 5 years
* Lung volume reduction surgery in previous 12 months
* Nocturnal positive pressure for sleep apnea
* Other inclusion and exclusion criteria will be evaluated at the first study visit.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2006-03; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Peripheral airway resistance measured by IOS

SECONDARY OUTCOMES:
Airway wall thickness measured by CT scans

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- United States (4):
  - GSK Investigational Site, Absecon, New Jersey
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
- Chile (2):
  - GSK Investigational Site, Valparaíso, Región de Valparaíso
  - GSK Investigational Site, Santiago, Región Metro de Santiago
- GSK Investigational Site, Tartu, Estonia
- Russia (3):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Nizhnekamsk

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Kreindler JL, Watkins ML, Lettis S, Tal-Singer R, Locantore N. Effect of inhaled corticosteroids on blood eosinophil count in steroid-naive patients with COPD. BMJ Open Respir Res. 2016 Sep 8;3(1):e000151. doi: 10.1136/bmjresp-2016-000151. eCollection 2016. PMID 27651909
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: SCO104925 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: SCO104925 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: SCO104925 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: SCO104925 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: SCO104925 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: SCO104925 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: SCO104925 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register